CLINICAL TRIAL: NCT00903435
Title: Quantitative Studies of Urinary Bladder Sensation
Status: Completed | Type: Observational
Sponsor: Timothy Ness, MD (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Timothy Ness, MD, M.D., Ph.D., University of Alabama at Birmingham
Organization: University of Alabama at Birmingham (Other)
Other Study IDs: F060505003; 3R01DK051413-11S1 (NIH)
Record Dates: First submitted 2009-04-23; First posted 2009-05-18 (Estimated); Last update posted 2011-12-01 (Estimated); Status verified 2011-11

CONDITIONS: Interstitial Cystitis
Keywords: Cystitis; Urinary; Bladder
MeSH Terms: conditions — Cystitis, Interstitial; Cystitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Quantitative Sensory Testing and Stimulus — No therapeutic intervention will be given. Quantitative Sensory Testing, thermal/mechanical/ischemic stimulus will be performed.

SUMMARY:
The purpose of this study is to determine whether more than one subpopulation exists of patients with the diagnosis of Interstitial Cystitis (IC) based on sensory testing and to determine if subjects with IC have normal counterirritation-related modulatory systems.

DETAILED DESCRIPTION:
To determine whether more than one subpopulation exists of patients with the diagnosis of Interstitial Cystitis (IC) based on sensory testing and to determine if subjects with IC have normal counterirritation-related modulatory systems. Previous studies by the PI suggest that two populations of subjects are present in the IC population but a larger number of subjects with IC would need to be tested in order to determine if this were indeed true. Other studies have demonstrated that counterirritation-related effects are absent in several chronic pain populations including fibromyalgia and chronic headaches. Identification of a subset of IC patients or the identification of a failure of counterirritation-related effects may predict responses to therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to read and speak English
* 19 years or older
* IC Diagnosis

Exclusion Criteria:

* Over 65 years old
* Pregnant
* Children younger than 19
* Significant cardiac disease

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Non-healthy subjects will be recruited from Kirklin Clinic Urology Clinic and Pain Treatment Center. Healthy subjects will be recruited via advertisements.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2007-05; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
The study proposes to examine the sensations that are produced by warming the skin, poking the skin, pressure on the muscles or by applying a blood pressure cuff. | One and a half to two hours

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Ness, M.D., Ph.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Kirklin Clinic, Birmingham, Alabama, United States